CLINICAL TRIAL: NCT01140841
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Dose-Escalation Study of Safety and Tolerability of Oromucosal Fipamezole ODT in Adult Subjects With Parkinson's Disease Who Are Receiving Levodopa
Brief Title: A Study of Safety and Tolerability of Fipamezole in Adult Subjects With Parkinson's Disease Who Are Receiving Levodopa
Acronym: Fipamezole
Status: Completed | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BVF-025-101
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Parkinson's Disease
Keywords: Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fipamezole ODT
  Interventions: Drug: Fipamezole ODT
- Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fipamezole ODT — Subjects take three daily doses of Fipamezole ODT, with each dose escalating from 30 to 60, 90, 120, 150 and up to 180 mg over 8 weeks.
  Groups: Fipamezole ODT
Drug: Placebo — 1 to 2 tablets three times per day to be taken according to the same schedule as the active study drug.
  Groups: Placebo

SUMMARY:
The purpose of this clinical trial is to determine the maximum tolerated dose of Fipamezole in adult patients with Parkinson's disease who are receiving levodopa.

DETAILED DESCRIPTION:
Parkinson's Disease is the second most common neurodegenerative disorder worldwide. While treatment with dopaminergic agents like levodopa, the mainstay of treatment, is effective in the early phases of the disease, their benefits decrease with disease progression, and problems such as dyskinesia and on-off phenomenon begin to manifest. In this study, fipamezole, a new antagonist of an adrenergic receptor, is being investigated to better understand the safety and side-effect profile in patients with Parkinson's Disease.

The sampling method used was simple random sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a man or woman between 30 and 75 years of age, inclusive, with intact oral mucosa at Screening (Visit 1) and Randomization (Visit 2).
2. Subject has a diagnosis of idiopathic Parkinson's disease defined according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis criteria.
3. Subject has been receiving a stable regimen of at least three daily administrations of levodopa (with a peripheral dopa decarboxylase inhibitor), with no dose changes for at least 4 weeks prior to Randomization (Visit 2).
4. Subject is rated at stage 2 to 4 on the Hoehn and Yahr scale.
5. If currently taking other medications (other than levodopa), subject must be on a stable regimen, defined as no dose changes for at least 1 month prior to Randomization (Visit 2).
6. Subject demonstrates the ability to comprehend the study procedures and provide informed consent.
7. Female subjects must be either postmenopausal for at least 1 year or surgically sterilized at least 3 months prior to Randomization (Visit 2). Male subjects must either be sterile or willing to use 2 approved methods of contraception when engaged in sexual intercourse with a female partner from Randomization (Visit 2) until 30 days after the last dose of study drug.
8. Subject has an upper arm circumference of not less than 24 cm and not more than 42 cm for both arms.

Exclusion Criteria:

1. Subject participated in an investigational medication study within the 3 months prior to Randomization (Visit 2).
2. Subject has immediate family members who are site Investigators or sponsor employees.
3. Subject has a history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
4. Subject has impaired renal function (defined as a creatinine level of ≥ 1.5 times the upper limit of normal) at Screening (Visit 1).
5. Subject has impaired hepatic function (defined as SGOT/AST or SGPT/ALT levels ≥ 1.5 times the upper limit of normal) at Screening (Visit 1).
6. Subject has second- or third-degree atrioventricular block or sick sinus syndrome, atrial fibrillation, atrial flutter, severe or unstable angina, congestive heart failure, or myocardial infarction within 3 months of the screening visit or a significant ECG abnormality, including a QRS > 110 msec, a PR interval > 230 msec, a QTc ≥ 450 msec for male subjects, or a QTc ≥ 470 msec for female subjects.
7. Subject has a history of risk factors for Torsades de Pointes, including unexplained syncope, known long QT syndrome, or a clinically significant abnormal laboratory assessment such as hypokalemia, hypercalcemia, or hypomagnesemia. Subjects with a family history of long QT syndrome or Brugada syndrome will also be excluded.
8. Subject is at immediate risk of requiring hospitalization.
9. Subject has significant tremor or dyskinesia which, in the opinion of the Investigator, might interfere with reliable assessment of continuous Holter ECG and ABPM.
10. Subject has, in the opinion of the Investigator, a clinically important abnormality on his/her physical examination, electrocardiography, vital sign measurements, or laboratory assessment.
11. Subject is being treated with a disallowed medication that cannot be discontinued prior to Randomization (Visit 2) (See Table 6).
12. Subject has a current diagnosis of substance abuse or history of alcohol or drug abuse in the past 2 years prior to Screening (Visit 1).
13. Subject has positive findings on urine drug screen at Screening (Visit 1).
14. Subject has an allergy to fipamezole or its excipients.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease on stable regimen of levodopa
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose (MTD) of Fipamezole orally disintegrating tablets (ODT) in adult patients with Parkinson's disease. | Days -28 to 56

SECONDARY OUTCOMES:
To assess cardiovascular safety of ascending doses of Fipamezole ODT in adult patients with Parkinson's disease. | Days -28 to 56
To evaluate pharmacokinetics (PK) of ascending doses of Fipamezole ODT in adult patients with Parkinson's disease. | Days -28 to 56
To assess incidence and severity of Adverse Events | Days -28 to 63

CONTACTS AND LOCATIONS:
Overall Officials: Karen Briegs, Study Director — Biovail Technologies, Ltd.
Locations (4):
- United States (4):
  - CNS Network, Inc., Torrance, California
  - Quest Research Institute, Bingham Farms, Michigan
  - Clinical Research Integrity Worldwide LLC, Willingboro, New Jersey
  - Duke University Medical Center, Durham, North Carolina